CLINICAL TRIAL: NCT06856668
Title: A Megastudy of Single-Session Interventions to Challenge Depression in American Adults
Brief Title: A Megastudy of Single-Session Interventions for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica Schleider, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU 00220193; 5T32MH115882-07 (NIH)
Record Dates: First submitted 2025-01-27; First posted 2025-03-04 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Depression - Major Depressive Disorder
Keywords: single-session intervention; depression; megastudy; digital mental health intervention; experiment; randomized clinical trial
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: All intervention conditions will be allocated approximately the same number of participants, while the control condition will be allocated three times that number.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Passive control (All About Trout) (Other): The passive control condition aims to hold one's attention for 8-10 minutes without influencing depressive symptoms or mood (a three-minute video, multiple-choice questions, two-minute reading passage, three-minute writing exercise, all about trout).
  Interventions: Behavioral: All about Trout
- Behavioral Activation (Action Brings Change Project) (Active Comparator): A behavioral activation SSI where users learn about negative thought spirals, share advice with an imagined peer, and create an "action plan" of helpful activities to engage in in the future.
  Interventions: Behavioral: Behavioral Activation (Action Brings Change Project 10-Minute Version)
- SSI 1: Mindful Acceptance (Experimental): A clinical psychologist explains a few ways to use mindful acceptance to deal with difficult thoughts and feelings.
  Interventions: Behavioral: Mindful Acceptance
- SSI 2: Moral Elevation (Experimental): Users learn about moral elevation, then watch a touching video where a man does good deeds for people in his community. Finally, they plan a positive action they can take to help others in their own life.
  Interventions: Behavioral: Moral Elevation
- SSI 3: Mindful Attention Skills (Experimental): A series of videos teach mindfulness skills: how to release thoughts and re-evaluate.
  Interventions: Behavioral: Mindful Attention Skills
- SSI 4: 5 Habits to Beat Depression (Experimental): A clinical psychologist and science communicator describes his top 5 one-minute habits to beat depression.
  Interventions: Behavioral: 5 Habits to Beat Depression
- SSI 5: Interactive Cognitive Reappraisal (Experimental): An interactive SSI where participants learn how to reframe negative thoughts.
  Interventions: Behavioral: Interactive Cognitive Reappraisal
- SSI 6: Expressive Writing (AI-supported) (Experimental): Participants describe a persistent negative thought they struggle with and a large language model system helps them to consider a story in which someone learns to overcome that thought.
  Interventions: Behavioral: Expressive Writing (AI-supported)
- SSI 7: Inner Child Healing Walk (Experimental): An interactive journey to reconnect and heal one's inner child through breathing exercises, positive affirmations, and supportive animal companions.
  Interventions: Behavioral: Inner Child Healing Walk
- SSI 8: Savoring Strategies (Experimental): An SSI introducing savoring strategies to improve mood.
  Interventions: Behavioral: Savoring Strategies
- SSI 9: Personalized Intervention Recommender (Experimental): Identifies the kinds of depression one struggles most with and offers a personalized recommendation for future depression support options.
  Interventions: Behavioral: Personalized Intervention Recommender
- SSI 10: Dialectical Behavioral Therapy Skills (Experimental): Presents videos from dialectical behavioral therapy on various ways to control negative emotions.
  Interventions: Behavioral: Dialectical Behavioral Therapy Skills
- SSI 11: Reframing Negative Thoughts (Experimental): An audio-only program in which users are guided to reflect on how they might challenge negative automatic thoughts and beliefs they struggle with.
  Interventions: Behavioral: Reframing Negative Thoughts

INTERVENTIONS:
Behavioral: Behavioral Activation (Action Brings Change Project 10-Minute Version) — A behavioral activation SSI where users learn about negative thought spirals, give advice to an imagined peer, then create an "action plan" of helpful activities to do in the near future. This is a shorter version of the original 15-minute Action Brings Change SSI.
  Other Names: ABC Project
  Arms: Behavioral Activation (Action Brings Change Project)
Behavioral: Mindful Acceptance — A clinical psychologist explains a few ways to use mindful acceptance to deal with difficult thoughts and feelings.
  Arms: SSI 1: Mindful Acceptance
Behavioral: Moral Elevation — Users learn about moral elevation, then watch a touching video where a man does good deeds for people in his community (originally a Thai life insurance advertisement). Finally, they plan a positive action they can take to help others in their own life.
  Arms: SSI 2: Moral Elevation
Behavioral: Mindful Attention Skills — A series of videos teach mindfulness skills: how to release thoughts and re-evaluate negative interpretations.
  Arms: SSI 3: Mindful Attention Skills
Behavioral: 5 Habits to Beat Depression — A clinical psychologist and science communicator describes his top 5 one-minute habits to beat depression.
  Arms: SSI 4: 5 Habits to Beat Depression
Behavioral: Interactive Cognitive Reappraisal — An interactive SSI where participants learn how to reframe negative thoughts
  Arms: SSI 5: Interactive Cognitive Reappraisal
Behavioral: Expressive Writing (AI-supported) — Participants describe a negative thought they struggle with and an LLM helps them to consider a story in which a peer overcomes that thought.
  Arms: SSI 6: Expressive Writing (AI-supported)
Behavioral: Inner Child Healing Walk — An interactive journey to reconnect and heal one's inner child through breathing exercises, positive affirmations, and supportive animal companions.
  Arms: SSI 7: Inner Child Healing Walk
Behavioral: Savoring Strategies — An SSI introducing savoring strategies to improve mood.
  Arms: SSI 8: Savoring Strategies
Behavioral: Personalized Intervention Recommender — Identifies the kinds of depression one struggles most with and offers a personalized recommendation for future depression support options
  Arms: SSI 9: Personalized Intervention Recommender
Behavioral: Dialectical Behavioral Therapy Skills — Presents videos from dialectical behavioral therapy on various ways to control negative emotions.
  Arms: SSI 10: Dialectical Behavioral Therapy Skills
Behavioral: All about Trout — An 8-10 minute educational program with information and interactive exercises about trout fish. Intended to capture one's attention and require some effort, while minimizing influence on depressive symptoms.
  Other Names: Passive control activity
  Arms: Passive control (All About Trout)
Behavioral: Reframing Negative Thoughts — An audio-only program in which users are guided to reflect on how they might challenge negative automatic thoughts and beliefs they struggle with.
  Arms: SSI 11: Reframing Negative Thoughts

SUMMARY:
This project aims to learn if new kinds of digital single-session interventions (SSIs) for depression could be effective for American adults. Many existing SSIs are delivered in a simple text-based format. However, it might be that different kinds of SSIs (in terms of both content and style) also have potential for scalable impact. Specifically, this study will investigate the effectiveness of 11 innovative SSIs by comparing them to a passive control and to an existing SSI with established efficacy.

ELIGIBILITY:
Inclusion criteria:

* At least 18 years old
* Able to read and write fluently in English
* Have enough access to the internet to complete two sessions over four weeks
* Score at least 10 on the PHQ-9 screen (suggesting moderate depression; Kroenke et al., 2001)
* Pass the bot check during the screening survey

All participants who are randomized to an experimental condition (and therefore completed all baseline measures) will be included in analyses, except for participants who indicate at the end of either the baseline or week 4 session that they did not participate in the study seriously. Researchers will only keep data from the first survey session a participant begins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7505 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-06-24 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire-9 at week 4 (PHQ-9; Kroenke et al., 2001) | Baseline to week 4
  The Patient Health Questionnaire-9 is a validated and self-administered measure to assess depression symptom severity in the general population. Participants are asked to rate how often they are bothered by 9 items (e.g., Poor appetite or overeating) on a scale of 0 (Not at all) to 3 (Nearly every day). Total score can range from 0 to 27, with higher scores indicating higher symptom severity.

SECONDARY OUTCOMES:
Change in Beck Hopelessness Scale at immediate post-intervention (BHS-4; Perczel Forintos et al., 2013) | Baseline to immediate post-intervention
  Beck Hopelessness Scale-4 is the 4-item version of the 20-item Beck Hopelessness scale (Beck et al. 1974). Participants will be asked to rate 4 items assessing different aspects of hopelessness (e.g., My future seems dark to me) on a scale of 0 (Absolutely disagree) to 3 (Absolutely agree). Total score can range between 0 to 12 with higher scores indicating higher hopelessness.
Change in Beck Hopelessness Scale at week 4 (BHS-4; Perczel Forintos et al., 2013) | Baseline to week 4
  Beck Hopelessness Scale-4 is the 4-item version of the 20-item Beck Hopelessness scale (Beck et al. 1974). Participants will be asked to rate 4 items assessing different aspects of hopelessness (e.g., My future seems dark to me) on a scale of 0 (Absolutely disagree) to 3 (Absolutely agree). Total score can range between 0 to 12 with higher scores indicating higher hopelessness.
Change in Pathways Subscale of the State Hope Scale at immediate post-intervention (Snyder et al., 1996) | Baseline to immediate post-intervention
  The "pathways" subscale reflects perceived success in meeting one's goals (eg, "At this time, I am meeting the goals I have set for myself"). Immediately pre- and post-intervention, participants rate each of 3 statements to reflect how they felt about themselves right now on an 8-point Likert scale.
Change in Pathways Subscale of the State Hope Scale at week 4 (Snyder et al., 1996) | Baseline to week 4
  The "pathways" subscale reflects perceived success in meeting one's goals (eg, "At this time, I am meeting the goals I have set for myself"). Immediately pre- and post-intervention, participants rate each of 3 statements to reflect how they felt about themselves right now on an 8-point Likert scale.
Change in Readiness for Change at immediate post-intervention | Baseline to immediate post-intervention
  To evaluate readiness for change at pre-test, post-test, and follow-up, participants will be asked two questions regarding making changes to reduce their feelings of depression: 1. "How important is making changes toward overcoming depression to you right now?" (1-4, Not at all- Extremely important) and 2. "How confident are you about making changes toward overcoming depression?" (1-4, Not at all- Extremely confident).
Change in Readiness for Change at week 4 | Baseline to week 4
  To evaluate readiness for change at pre-test, post-test, and follow-up, participants will be asked two questions regarding making changes to reduce their feelings of depression: 1. "How important is making changes toward overcoming depression to you right now?" (1-4, Not at all- Extremely important) and 2. "How confident are you about making changes toward overcoming depression?" (1-4, Not at all- Extremely confident).
Change in Depression Expectancies for Change at immediate post-intervention (Eddington et al., 2014) | Baseline to immediate post-intervention
  To evaluate how much people expect to be able to change their symptoms of depression, participants will respond to the three items with the highest item-total correlation from the Depression Expectancies for Change scale (Eddington et al., 2014). These are rated on a 5-point likert scale from 1 (strongly disagree) to 5 (strongly agree). Items 1 and 2 are reverse-coded.
Change in Depression Expectancies for Change at week 4 (Eddington et al., 2014) | Baseline to week 4
  To evaluate how much people expect to be able to change their symptoms of depression, participants will be asked to respond to three items with the highest item-total correlation from the Depression Expectancies for Change scale (Eddington et al., 2014). These are rated on a 5-point likert scale from 1 (strongly disagree) to 5 (strongly agree). Items 1 and 2 are reverse-coded.
Change in Frequency of Actions and Thoughts Scale at immediate post-intervention (FATS; Terides et al., 2016). | Baseline to immediate post-intervention
  A 12-item measure of adaptive thoughts and behaviors, improvement in which might be a target of psychotherapy. Range 0-48 with higher scores indicating greater frequency of adaptive thoughts and behaviors.
Change in Frequency of Actions and Thoughts Scale at week 4 (FATS; Terides et al., 2016). | Baseline to week 4
  A 12-item measure of adaptive thoughts and behaviors, improvement in which might be a target of psychotherapy. Range 0-48 with higher scores indicating greater frequency of adaptive thoughts and behaviors.
Credibility and Expectancy Questionnaire at immediate post-intervention (CEQ; Devilly & Borkovec; 2000) | immediate post-intervention
  A 6-item measure of user-perceived intervention appeal and efficacy. Range 6-54 with higher scores indicating higher user-perceived intervention appeal and efficacy.
Insight Experience at immediate post-intervention | immediate post-intervention
  Participants will be asked two questions about users' insight experiences, with the following text:
  The next question will ask if you experienced an "Aha! Moment".
  You can think of this experience as a miniature 'Eureka moment'. You might even feel an internal sense of "Aha!," or you might think to yourself, "of course!," "that was so obvious". Not experiencing an Aha! moment might feel like nothing much at all.
  1. Did something in the program make you experience an Aha! Moment? (No 0 / Yes 1)
  2. How significant did you feel this Aha! Moment was? In other words, how much do you feel it will have a lasting impact on you? 1 (not at all significant) - 5 (very significant)
Insight Experience at week four | week 4
  Participants will be asked three questions about whether they had an insight experience during the SSI, with the following text:
  The next question will ask if you experienced an "Aha! Moment".
  You can think of this experience as a miniature 'Eureka moment'. You might even feel an internal sense of "Aha!," or you might think to yourself, "of course!," "that was so obvious". Not experiencing an Aha! moment might feel like nothing much at all.
  1. Did something in the program make you experience an Aha! Moment *that you still remember today*? (No 0 / Yes 1)
  2. How significant did you feel this Aha! Moment was? In other words, how much do you feel it will have a lasting impact on you? 1 (not at all significant) - 5 (very significant)
  3. How much has the Aha! Moment you experienced changed the way that you think or act? 1 (not at all) - 5 (a great deal)
Star rating at immediate post-intervention | immediate post-intervention
  Participants rate the overall quality of the program they completed from 1-5 stars, with 5 being the best. (5 stars to fill in, discrete 1-5)
Star rating at week 4 | week 4
  Participants rate the overall quality of the program they completed from 1-5 stars, with 5 being the best. (5 stars to fill in, discrete 1-5)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Medical Social Sciences, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers will share all non-identifiable individual participant data (IPD) from the study.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The IPD and supporting information will be available by July 30, 2025, with no end date.
Access Criteria: The IPD will be publicly available online via the study open science framework (OSF) page (https://osf.io/agvh6)
URL: https://osf.io/agvh6

REFERENCES:
- [Background] Eddington KM, Dozois DJ, Backs-Dermott BJ. Evaluation of the internal consistency, factor structure, and validity of the Depression Change Expectancy Scale. Assessment. 2014 Oct;21(5):607-17. doi: 10.1177/1073191113517929. Epub 2013 Dec 30. PMID 24379447
- [Background] Terides MD, Dear BF, Karin E, Jones MP, Gandy M, Fogliati VJ, Kayrouz R, Staples LG, Titov N. The frequency of actions and thoughts scale: development and psychometric validation of a measure of adaptive behaviours and cognitions. Cogn Behav Ther. 2016 Apr;45(3):196-216. doi: 10.1080/16506073.2016.1149876. Epub 2016 Feb 29. PMID 26926484
- [Background] Snyder CR, Sympson SC, Ybasco FC, Borders TF, Babyak MA, Higgins RL. Development and validation of the State Hope Scale. J Pers Soc Psychol. 1996 Feb;70(2):321-35. doi: 10.1037//0022-3514.70.2.321. PMID 8636885
- [Background] Perczel Forintos D, Rozsa S, Pilling J, Kopp M. Proposal for a short version of the Beck Hopelessness Scale based on a national representative survey in Hungary. Community Ment Health J. 2013 Dec;49(6):822-30. doi: 10.1007/s10597-013-9619-1. Epub 2013 Jun 12. PMID 23756722
- [Background] Laukkonen RE, Kaveladze BT, Tangen JM, Schooler JW. The dark side of Eureka: Artificially induced Aha moments make facts feel true. Cognition. 2020 Mar;196:104122. doi: 10.1016/j.cognition.2019.104122. Epub 2019 Nov 20. PMID 31759277
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Goodman E, Adler NE, Kawachi I, Frazier AL, Huang B, Colditz GA. Adolescents' perceptions of social status: development and evaluation of a new indicator. Pediatrics. 2001 Aug;108(2):E31. doi: 10.1542/peds.108.2.e31. PMID 11483841
- [Background] Devilly GJ, Borkovec TD. Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry. 2000 Jun;31(2):73-86. doi: 10.1016/s0005-7916(00)00012-4. PMID 11132119
- [Background] Beck AT, Weissman A, Lester D, Trexler L. The measurement of pessimism: the hopelessness scale. J Consult Clin Psychol. 1974 Dec;42(6):861-5. doi: 10.1037/h0037562. No abstract available. PMID 4436473
- [Derived] Kaveladze B, Voelkel J, Stagnaro M, Huang M, Smock A, Sullivan E, Xu Y, McCall M, Zapata JP, Ishtiaque S, Bhattacharjee A, Georgieva I, Hernandez-Ramos R, Huber K, Jennings J, Kirk A, Kornfield R, Knowles R, Lind M, Liu M, Liut M, Mariakakis A, Mattu A, McGuire A, Meyerhoff J, Mrazek A, Mrazek M, Mohr D, Morris R, Mosunic C, Nip H, Olson-Urtecho A, Podell J, Ransom D, Rizvi S, Southward M, Stoeckl SE, Taylor M, Texter A, Trotter A, Tower C, Williams J, Woodson E, Wislocki K, Protzko J, Lorenzo-Luaces L, Schueller S, Nock M, Schleider J. A Crowdsourced Megastudy of 12 Digital Single-Session Interventions for Depression in American Adults. Res Sq [Preprint]. 2025 Aug 25:rs.3.rs-7236847. doi: 10.21203/rs.3.rs-7236847/v1. PMID 40909806
- See also: Study Open Science Framework page with data and more information — https://osf.io/agvh6

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT06856668/Prot_SAP_ICF_001.pdf